CLINICAL TRIAL: NCT06623227
Title: Randomized, Placebo-controlled, Double-blind Study of Increasing Total Antioxidant Capacity with Vitamin E and C in Two Cohorts of Patients with Autism Spectrum Disorders
Brief Title: Effect of Increasing Total Antioxidant Capacity in Autism Spectrum Disorder
Acronym: TACASD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rinvil Renaldi (Other)
Collaborators: University of Modena and Reggio Emilia (Other); Indonesia University (Other); RSUP Dr. Wahidin Sudirohusodo (Other)
Responsible Party: Sponsor-Investigator, Rinvil Renaldi, MD, Child and Adolescent Psychiatrist, Hasanuddin University
Organization: Hasanuddin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAC_Study_ASD
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Total antioxidant capacity; Autism; Clinical symptoms; Aberrant behavior; Quality of life; Vitamin E; Vitamin C
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Vitamin E

STUDY DESIGN:
Intervention Model Description: Each patients treated with Risperidone and Behavior Therapy as maintanence therapy will divided into a controled group which receive plasebo and the other as intervention group which received Vitamin E (150-200 IU/d) and C (100-200 mg/d) for 3 months. Patients are assessed at T0, T6 and T12 wk. Administration of active compound and placebo is in double-blind.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, all care providers, investigators and outcome assessors are blind to treatment status, as well as patients and family. Three investigators, who have no direct contact with patients and families, are responsible for managing the study procedures or treatments. Another investigator, who is not involved in assessing the outcomes, interacts with families to answer any questions regarding the trial or medical issues. This investigator also ensures that the outcome assessors are not influenced by any contact with families between the assessment periods (0, 6, and 12 weeks). Families are asked to refrain from discussing their experiences and the trial outcomes on social media.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ASD Placebo (Active Comparator): If the age is up to 4 years old:
  • Risperidone (0.02-0.06 mg/KgBW) and Behavior Therapy as maintenance therapy and Capsule Placebo.
  If age is above 4 years old:
  • Risperidone (0.02-0.06 mg/KgBW) and Behavior Therapy as maintenance therapy and Capsule Placebo.
  Interventions: Dietary Supplement: Placebo
- ASD Active compound (Experimental): If the age is up to 4 years old:
  • Risperidone (0.02-0.06 mg/KgBW) and Behavior Therapy as maintenance therapy and Capsul containing Vitamin E 150 IU and Vitamin C 100 mg.
  If age is above 4 years old:
  • Risperidone (0.02-0.06 mg/KgBW) and Behavior Therapy as maintenance therapy and Capsul containing Vitamin E 200 IU and Vitamin C 200 mg.
  Interventions: Dietary Supplement: Vitamin E and C

INTERVENTIONS:
Dietary Supplement: Placebo — Capsule contains substances that are safe, non-active, and commonly used in pharmaceuticals (microcrystalline cellulose) with an appropriate coloring dye and in the active arms, Vitamin E and C. Capsules can be opened and the content drunk or chewed, if children have difficulties with swallowing capsules
  Arms: ASD Placebo
Dietary Supplement: Vitamin E and C — Capsule Vitamin E (Natural Vitamin E, d-alpha tocopherol) 150 IU or 200 IU containing also Vitamin C 100 mg or 200 mg b.id depending on age. Capsules can be opened and the content drunk or chewed, if children have difficulties with swallowing capsules
  Arms: ASD Active compound

SUMMARY:
This double-blind, randomized, controlled trial (RCT) has the aim to evaluating the effectiveness of increasing Total Antioxidant Capacity (TAC) as add-on intervention in two cohorts of patients with Autism Spectrum Disorder (ASD) who have received Risperidone (0.02-0.06 mg/KgBW) and Behavior Therapy as maintenance therapy. Both groups will receive placebo pill or Vitamin E and C pill using randomization. Clinical Symptoms, Aberrant Behavior and Quality of Life in Children with ASD will be assessed after 12 weeks of treatment in this study. Primary outcome measures of efficacy is Aberrant Behavior Checklist- Irritability (ABC-Irritability) and Secondary outcome measures include Childhood Autism Rating Scale (CARS), Clinical Global Impression Scale - Improvement (CGI-I), The PedsQL and The WHOQOL BREF.

DETAILED DESCRIPTION:
The continuation of ASD throughout life makes all efforts to optimize the abilities of children with ASD as early as possible so that their quality of life becomes better important. Management to improve current symptoms and overcome aberrant behavior in children with ASD generally focuses on behavioral intervention, psychotherapy and even pharmacotherapy, but the results are not satisfactory because it takes time, is expensive and unexpected side effects often occur after administering pharmacotherapy. On the other hand, research related to the role of oxidative stress has suggested a potential relationship between oxidative stress and autism pathophysiology that is not correlated with age and the underlying pathogenesis, but damage caused by oxidative stress will exacerbate dysfunction in children with ASD through chronic inflammatory responses, DNA and protein damage and mitochondrial superoxide production. Oxidative stress will influence the clinical symptoms and pathogenesis of ASD. Therefore, efforts to control the balance of oxidative stress to improve symptoms and neuropsychological deficits in patients with ASD are important. Lack of antioxidant capacity in children with ASD to neutralize and remove oxidants has been associated with the severity of clinical symptoms and aberrant behavior in children with ASD. Therefore, efforts to increase antioxidant capacity through providing antioxidants can offer a new strategy for dealing with accompanying symptoms in children with ASD.

Vitamin E and Vitamin C are non-enzymatic antioxidants which function to strengthen the work of enzymatic antioxidants in the oxidant-elimination, oxidation-reduction cycle process that occurs in the brain. Its includes in group of antioxidants which also referred as chain breaking. When used together with vitamin C which can function as a water-soluble antioxidant and other enzyme cofactors, reduced vitamin C can directly regenerate vitamin E which simultaneously undergoes oxidation to become ascorbate. Therefore, the use of vitamin C will be more effective when used together with vitamin E. Research has shown that administration with antioxidants such as vitamin E and vitamin C has a good effect on clinical symptoms and behavior in children with ASD.

In this randomized controlled trial (RCT), patients with Autism Spectrum Disorder (ASD) who have received Risperidone and Behavior Therapy as maintenance therapy will be randomly assigned to receive either a placebo or a combination of Vitamins E (150-200 IU per day) and C (100-200 mg per day) for a duration of 3 months. This study was designed to verify whether increasing the TAC using Vitamin E and C improves clinical symptoms, aberrant behaviors, and quality of life in children with ASD.

This study shall include 50 patients with ASD, aged 3-9 years old. The study design of this RCT was balanced to all of patients treated with maintenance therapy as usual, so that half of the patients will receive placebo, and the remaining half will receive Vitamin E and C during 3 months. The purpose is to observe whether the increase of TAC could improve the clinical symptoms, aberrant behavior and quality of life in ASD patients. In addition to clinical and psychometric parameters, TAC will be measured at baseline, after 6 weeks and 12 weeks, by collecting 30-60 ml of fresh urine, a general urinalysis examination to rule out acute urinary tract infections, The TAC examination is carried out when the urine pH is normal and measurement with a calorimetric kit with enzyme method, ABTS.

ELIGIBILITY:
Inclusion Criteria:

1. Both parents or a legally authorized patient representative (LAR) must provide written informed consent. The parents and guardian must be able to understand and comply with the experimental protocol with a minimum of junior high school education.
2. Parents earn no less than IDR 3,434,298 (South Sulawesi Province Minimum Wage for 2024).
3. Subjects of both sexes, aged between 3-9 years old, may be included in the study.
4. The subject must meet DSM-5 criteria for a primary diagnosis of Autism.
5. Patients treated with Risperidone (0.02-0.06 mg/KgBW) are enrolled only if the treatment and dosage of these drugs has been constant for at least 2 months prior to enrollment in the trial and is kept constant throughout the 3-month duration of the trial.
6. Patients undergoing any kind of behavioral intervention must have must have underwent the intervention at least 2 sessions prior to enrollment and the intervention must remain unchanged throughout the 3-month duration of the trial.
7. Baseline Clinical Global Impression - Severity (CGI-S) score below 7.
8. The patient is able to swallow the capsule or his/her parents are available to open it and administer immediately its content in a small quantity of juice or soft-drink.

Exclusion Criteria:

1. Patients with organic disease and/or congenital malformation including known genetic syndromes for example, Rett syndrome, fragile-X syndrome, and Down Syndrome etc.).
2. Patients with autism secondary to epileptic encephalopathy or with idiopathic autism co-morbid with seizures more frequent than one episode every 6 months despite ongoing anti epileptic drug therapy.
3. Patients treated with anticoagulants.
4. Patients with serious medical illnesses (chronic renal disease, severe liver disease, cardiovascular disorders, malignant tumors, HIV infection).
5. Patients with a history of acute cerebrovascular episodes.
6. Patients with a history of stomach bleeding or active peptic ulcer.
7. Patients with documented allergy, hypersensitivity or intolerance to one of the excipients of the experimental or comparative product.
8. Patients have been consuming other antioxidants.
9. Patients with active urinary tract infections.
10. Patients with poor compliance and or no control back to the Hospital.

Trial interruption criteria:

1. Patients whose medical conditions require starting treatment with anticoagulants.
2. Patients with severe medical conditions starting during the 3-month duration of the trial.
3. Patients who undergo a change in psychopharmacological or behavioral treatment during the 3-month duration of the trial.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-09-28 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist - Irritability (ABC-I) | At 0, 6 and 12 weeks duration of trial
  An instrument which is used by parents to measure aberrant behavior in children which consists of 15 assessment items with a scale of 0-3 to assess the level of severity. Score between 0-45 with interpretation if score <20, mild; 20-40 moderate; >40, severe irritability.

SECONDARY OUTCOMES:
Childhood Autism Rating Scale (CARS) | At 0, 6 and 12 weeks duration of trial
  CARS is an instrument for measuring the severity of signs and symptoms of ASD carried out by experienced clinicians. Score between 15-60 with interpretation if score <30, non-autistic; 30-36.5 mild to moderate autism; 37-60, severe autism.
Clinical Global Impression Scale- Improvement (CGI-I) | At 0, 6 and 12 weeks duration of trial
  a scale consisting of 7 assessment points used by clinicians to assess the severity of the patient's initial condition, patient improvement/worsening during follow-up and treatment side effects.
The Pediatric Quality of Life TM (The PedsQL) | At 0, 6 and 12 weeks duration of trial
  An instrument for assessing the quality of life in children related to health conditions, through self-assessment and/or parental observation, which is assessed based on conditions during the last 1 month.
WHOQOL-BREF | At 0, 6 and 12 weeks duration of trial
  An instrument for assessing parents' quality of life through self-assessment. The WHOQOL is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale.

CONTACTS AND LOCATIONS:
Overall Officials: Rinvil Renaldi, MD, Principal Investigator — Hasanuddin University
Locations (1):
- Doctoral Programme at Hasanuddin University, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Persico AM, Arango C, Buitelaar JK, Correll CU, Glennon JC, Hoekstra PJ, Moreno C, Vitiello B, Vorstman J, Zuddas A; European Child and Adolescent Clinical Psychopharmacology Network. Unmet needs in paediatric psychopharmacology: Present scenario and future perspectives. Eur Neuropsychopharmacol. 2015 Oct;25(10):1513-31. doi: 10.1016/j.euroneuro.2015.06.009. Epub 2015 Jun 20. PMID 26166453
- [Background] Adams JB, Audhya T, McDonough-Means S, Rubin RA, Quig D, Geis E, Gehn E, Loresto M, Mitchell J, Atwood S, Barnhouse S, Lee W. Effect of a vitamin/mineral supplement on children and adults with autism. BMC Pediatr. 2011 Dec 12;11:111. doi: 10.1186/1471-2431-11-111. PMID 22151477
- [Background] Zambrelli E, Lividini A, Spadavecchia S, Turner K, Canevini MP. Effects of Supplementation With Antioxidant Agents on Sleep in Autism Spectrum Disorder: A Review. Front Psychiatry. 2021 Jun 28;12:689277. doi: 10.3389/fpsyt.2021.689277. eCollection 2021. PMID 34262494
- [Background] Wang L, Wang B, Wu C, Wang J, Sun M. Autism Spectrum Disorder: Neurodevelopmental Risk Factors, Biological Mechanism, and Precision Therapy. Int J Mol Sci. 2023 Jan 17;24(3):1819. doi: 10.3390/ijms24031819. PMID 36768153
- [Background] Vargason T, Kruger U, Roth E, Delhey LM, Tippett M, Rose S, Bennuri SC, Slattery JC, Melnyk S, James SJ, Frye RE, Hahn J. Comparison of Three Clinical Trial Treatments for Autism Spectrum Disorder Through Multivariate Analysis of Changes in Metabolic Profiles and Adaptive Behavior. Front Cell Neurosci. 2018 Dec 19;12:503. doi: 10.3389/fncel.2018.00503. eCollection 2018. PMID 30618645
- [Background] Traber MG. Vitamin E: necessary nutrient for neural development and cognitive function. Proc Nutr Soc. 2021 Aug;80(3):319-326. doi: 10.1017/S0029665121000914. Epub 2021 Apr 26. PMID 33896432
- [Background] Teleanu DM, Niculescu AG, Lungu II, Radu CI, Vladacenco O, Roza E, Costachescu B, Grumezescu AM, Teleanu RI. An Overview of Oxidative Stress, Neuroinflammation, and Neurodegenerative Diseases. Int J Mol Sci. 2022 May 25;23(11):5938. doi: 10.3390/ijms23115938. PMID 35682615
- [Background] Silvestrini A, Meucci E, Ricerca BM, Mancini A. Total Antioxidant Capacity: Biochemical Aspects and Clinical Significance. Int J Mol Sci. 2023 Jul 1;24(13):10978. doi: 10.3390/ijms241310978. PMID 37446156
- [Background] Pangrazzi L, Balasco L, Bozzi Y. Natural Antioxidants: A Novel Therapeutic Approach to Autism Spectrum Disorders? Antioxidants (Basel). 2020 Nov 26;9(12):1186. doi: 10.3390/antiox9121186. PMID 33256243
- [Background] Hughes HK, R J Moreno, Ashwood P. Innate immune dysfunction and neuroinflammation in autism spectrum disorder (ASD). Brain Behav Immun. 2023 Feb;108:245-254. doi: 10.1016/j.bbi.2022.12.001. Epub 2022 Dec 6. PMID 36494048
- [Background] Liu X, Lin J, Zhang H, Khan NU, Zhang J, Tang X, Cao X, Shen L. Oxidative Stress in Autism Spectrum Disorder-Current Progress of Mechanisms and Biomarkers. Front Psychiatry. 2022 Mar 1;13:813304. doi: 10.3389/fpsyt.2022.813304. eCollection 2022. PMID 35299821
- [Background] Logan SL, Carpenter L, Leslie RS, Garrett-Mayer E, Hunt KJ, Charles J, Nicholas JS. Aberrant Behaviors and Co-occurring Conditions as Predictors of Psychotropic Polypharmacy among Children with Autism Spectrum Disorders. J Child Adolesc Psychopharmacol. 2015 May;25(4):323-36. doi: 10.1089/cap.2013.0119. Epub 2015 Apr 28. PMID 25919445
- [Background] Lee KH, Cha M, Lee BH. Neuroprotective Effect of Antioxidants in the Brain. Int J Mol Sci. 2020 Sep 28;21(19):7152. doi: 10.3390/ijms21197152. PMID 32998277
- [Background] Imataka G, Yui K, Shiko Y, Kawasaki Y, Sasaki H, Shiroki R, Yoshihara S. Urinary and Plasma Antioxidants in Behavioral Symptoms of Individuals With Autism Spectrum Disorder. Front Psychiatry. 2021 Sep 3;12:684445. doi: 10.3389/fpsyt.2021.684445. eCollection 2021. PMID 34539458
- [Background] Goel R, Hong JS, Findling RL, Ji NY. An update on pharmacotherapy of autism spectrum disorder in children and adolescents. Int Rev Psychiatry. 2018 Feb;30(1):78-95. doi: 10.1080/09540261.2018.1458706. Epub 2018 Apr 25. PMID 29693461
- [Background] Gabriele S, Sacco R, Persico AM. Blood serotonin levels in autism spectrum disorder: a systematic review and meta-analysis. Eur Neuropsychopharmacol. 2014 Jun;24(6):919-29. doi: 10.1016/j.euroneuro.2014.02.004. Epub 2014 Feb 19. PMID 24613076
- [Background] Frye RE. Mitochondrial Dysfunction in Autism Spectrum Disorder: Unique Abnormalities and Targeted Treatments. Semin Pediatr Neurol. 2020 Oct;35:100829. doi: 10.1016/j.spen.2020.100829. Epub 2020 Jun 23. PMID 32892956
- [Background] Doyle CA, McDougle CJ. Pharmacologic treatments for the behavioral symptoms associated with autism spectrum disorders across the lifespan. Dialogues Clin Neurosci. 2012 Sep;14(3):263-79. doi: 10.31887/DCNS.2012.14.3/cdoyle. PMID 23226952
- [Background] Cucinotta F, Ricciardello A, Turriziani L, Mancini A, Keller R, Sacco R, Persico AM. Efficacy and Safety of Q10 Ubiquinol With Vitamins B and E in Neurodevelopmental Disorders: A Retrospective Chart Review. Front Psychiatry. 2022 Mar 3;13:829516. doi: 10.3389/fpsyt.2022.829516. eCollection 2022. PMID 35308885
- [Background] Chauhan A, Chauhan V. Oxidative stress in autism. Pathophysiology. 2006 Aug;13(3):171-81. doi: 10.1016/j.pathophys.2006.05.007. Epub 2006 Jun 12. PMID 16766163
- [Background] Casanova MF, Frye RE, Gillberg C, Casanova EL. Editorial: Comorbidity and Autism Spectrum Disorder. Front Psychiatry. 2020 Nov 20;11:617395. doi: 10.3389/fpsyt.2020.617395. eCollection 2020. No abstract available. PMID 33329163
- [Background] Baraskewich J, von Ranson KM, McCrimmon A, McMorris CA. Feeding and eating problems in children and adolescents with autism: A scoping review. Autism. 2021 Aug;25(6):1505-1519. doi: 10.1177/1362361321995631. Epub 2021 Mar 2. PMID 33653157
- [Background] Aishworiya R, Valica T, Hagerman R, Restrepo B. An Update on Psychopharmacological Treatment of Autism Spectrum Disorder. Neurotherapeutics. 2022 Jan;19(1):248-262. doi: 10.1007/s13311-022-01183-1. Epub 2022 Jan 14. PMID 35029811
- [Background] Bjorklund G, Waly MI, Al-Farsi Y, Saad K, Dadar M, Rahman MM, Elhoufey A, Chirumbolo S, Jozwik-Pruska J, Kaluzna-Czaplinska J. The Role of Vitamins in Autism Spectrum Disorder: What Do We Know? J Mol Neurosci. 2019 Mar;67(3):373-387. doi: 10.1007/s12031-018-1237-5. Epub 2019 Jan 3. PMID 30607900